CLINICAL TRIAL: NCT04850911
Title: Reward Emotion Learning and Ketamine Study
Acronym: RELAKS
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: University of Oxford (Other)
Collaborators: Medical Research Council (Other Government); Johnson & Johnson Pharmaceutical Research & Development, L.L.C. (Industry)
Responsible Party: Principal Investigator, Catherine Harmer, Professor, University of Oxford
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Basic Science
Other Study IDs: RELAKS_HV
Record Dates: First submitted 2021-04-01; First posted 2021-04-20 (Actual); Last update posted 2023-03-28 (Actual); Status verified 2023-03

CONDITIONS: Depression; Major Depressive Disorder; Treatment Resistant Depression
Keywords: Ketamine; Learning; Memory; Habenula
MeSH Terms: conditions — Depression; Depressive Disorder, Major; Depressive Disorder, Treatment-Resistant | interventions — Ketamine

STUDY DESIGN:
Intervention Model Description: Participants will be assigned to receive either ketamine or placebo. Ketamine is not being administered for treatment purposes, the purpose is to understand the mechanisms underpinning its effects.
Who Masked: Participant, Investigator
Masking Description: All members of the study team will be blinded to the condition a participant is allocated to with the exception of the team member responsible for administering the drug/placebo.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Ketamine (Experimental): Participants in this arm will receive a single intravenous, antidepressant dose of ketamine hydrochloride (0.5mg/kg)
  Interventions: Drug: Ketamine Hydrochloride
- Placebo (Placebo Comparator): Participants in this arm will receive a single intravenous injection of an inactive placebo (0.9% sodium chloride).
  Interventions: Other: No intervention (placebo)

INTERVENTIONS:
Drug: Ketamine Hydrochloride — Ketamine is a high trapping NMDA receptor antagonist which has rapid and reliable antidepressant effects in patients with major depressive disorder (MDD) who have failed to respond to conventional monoaminergic agents.
  Arms: Ketamine
Other: No intervention (placebo) — Placebo injection (0.9% sodium chloride)
  Arms: Placebo

SUMMARY:
Ketamine's efficacy as an antidepressant is now well established yet the mechanisms underlying its antidepressant effect are yet to be fully described. Work in the animal literature and research in humans is suggestive of specific effects on anhedonia and memory reconsolidation. In this study the investigators will further explore the effects of ketamine on learning and memory as well as measuring the associated changes at neural level in a sample of healthy volunteers. Participants will be assigned to receive ketamine or placebo and complete a set of tasks which will allow the investigators to quantify the effect of ketamine on learning about reward and punishment and memory for learned reward associations 24 hours after ketamine infusion. This study will help the investigators to understand the basis of ketamine's antidepressant effects and aid the development of new treatments for depression.

ELIGIBILITY:
Inclusion Criteria:

* BMI between 18 and 30
* Participant is willing and able to give informed consent for participation in the study
* Sufficient knowledge of English language to understand and complete study tasks
* Willingness to refrain from driving, cycling, or operating heavy machinery, until the following morning or a restful sleep has occurred, whichever is later.
* Willingness to refrain from signing legal documents within 7 days after the infusion visit.
* Willingness to refrain from drinking alcohol for 3 days before the infusion visit and one day before any of the other visits throughout the study

Exclusion Criteria:

* Any current or past DSM-V significant psychiatric disorder including any psychotic, mood and anxiety and borderline personality disorders
* History of, or current medical conditions which in the opinion of the investigator may interfere with the safety of the participant or the scientific integrity of the study, including epilepsy/seizures, brain injury, hepatic or renal disease, severe gastro-intestinal problems, Central Nervous System (CNS) tumours, neurological conditions
* First-degree relative with a diagnosis of schizophrenia-spectrum or other psychotic disorder, or bipolar disorder
* History of unexplained hallucinations or impulse control problems (e.g. pathological gambling)
* Current or past history of heart rhythm disorders
* Clinically significant hypertension
* Increased intraocular pressure/glaucoma
* Current pregnancy (as determined by urine pregnancy test taken during Screening and Infusion Visits) or breastfeeding
* Clinically significant abnormal values for clinical chemistry (e.g. liver function tests), urine drug screen, blood pressure measurement and ECG. A participant with a clinical abnormality or parameters outside the reference range for the population being studied may be included only if the Investigator considers that the finding is unlikely to introduce additional risk factors and will not interfere with the study procedures
* Current or previous intake (last three months) of any medication that has a significant potential to affect mental functioning (e.g. benzodiazepines, antidepressants, neuroleptics etc.)
* Any intake of recreational drugs in the last 3 months (e.g. marijuana, ecstasy etc.)
* Lifetime recreational use of ketamine or phencyclidine
* Regular alcohol consumption of more than 14 units a week or excessive alcohol consumption up to three days before any of the in-person study visits
* Inability to abstain from alcohol for more than 1 week
* Regular smoker (> 5 cigarettes per day)
* Excessive caffeine user (> 6 caffeinated drinks per day)
* History of recurrent rashes or history of allergic reactions to relevant substances (ketamine treatment, placebo treatment)
* Previous participation in a study using the same or similar tasks
* Current participation in another study or participation in similar study within the last 6 months
* Participant is unlikely to comply with the clinical study protocol or is unsuitable for any other reason, in the opinion of the Investigator
* Claustrophobia
* Any implants (including dental implants) or pacemaker
* Tattoos above the chest
* Any other MRI contraindications outlined in FMRIB 7 Tesla scanning safety form

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 70 (Estimated)
Dates: Start 2021-08-25 (Actual); Primary Completion 2023-05 (Estimated); Study Completion 2023-05 (Estimated)

PRIMARY OUTCOMES:
Activation of the habenula during the Pavlovian conditioning task in response to the conditioned stimulus associated with pain stimuli and in response to the receipt of shock. | 24 hours after ketamine infusion
  Blood Oxygen Level Dependent (BOLD) signal in the habenula at the time of the shock-associated conditioned stimulus presentation and at the time of shock delivery.
Habenula response to the absence of expected reward and the receipt of an unexpected loss (i.e. a negative prediction error signal) in both the reward maximisation and loss minimisation tasks. | 24 hours after ketamine administration
  BOLD signal in the habenula at the time of outcome presentation in both the reward maximisation and loss minimisation tasks.
Preference for high-reward probability shapes learned after winning money (in the Wheel of Fortune draw) during the preference test. | +/- 24 hours after ketamine administration
  Proportion of choices where high-reward probability shapes are selected. This will be based on the difference between the perceived reward probability of shapes learned after the winning and losing of money (an area under the curve measure).

SECONDARY OUTCOMES:
Ventral striatum response to the expected reward and the omission an unexpected loss (i.e. a positive prediction error signal) in both the reward maximisation and loss minimisation tasks. | 24 hours after ketamine administration
  BOLD signal in the ventral striatum at the time of outcome presentation in both the reward maximisation and loss minimisation tasks.
Pupil dilation (measured by an eye tracker device) in response to decision values in the affective memory preference test. | 24 hours after ketamine administration
  Baseline corrected pupil dilation measured at the time of option presentation during each choice trial of the affective memory preference test.
Difference in pupil response to shapes learned after winning versus losing money. | 24 hours after ketamine administration
  Between groups comparison of pupil dilation in response to shapes learned after a loss and shapes learned after a win in Wheel of Fortune draw that induces experimental change in negative/positive affect.
Amount of money earned in the learning and memory task. | Final component completed 24 hours after ketamine administration before scanning
  Between groups comparison of the total amount of money earned during the learning and memory task.
Change in bio-behavioral measures of stress following laboratory induced stress administered. | 1-week after ketamine infusion
  Between groups comparison of salivary cortisol in response to Oxford Cognition Stress Task.
Change in bio-behavioral measures of stress following laboratory induced stress administered. | 1-week after ketamine infusion
  Between groups comparison of salivary alpha amylase in response to Oxford Cognition Stress Task.
Change in bio-behavioral measures of stress following laboratory induced stress administered. | 1-week after ketamine infusion
  Between groups comparison of heart rate in response to Oxford Cognition Stress Task.
Change in bio-behavioral measures of stress following laboratory induced stress administered. | 1-week after ketamine infusion
  Between groups comparison of visual analogue scale ratings in response to Oxford Cognition Stress Task.
Recognition of positive and negative facial expressions. | Immediately and 24 hours after ketamine infusion
  Recognition accuracy for positive and negative facial expressions
Recognition of positive and negative facial expressions. | Immediately and 24 hours after ketamine infusion
  Reaction time to recognise positive and negative facial expressions
Categorisation of emotional words. | 24 hours after ketamine infusion
  Accuracy of categorisation for positive and negative descriptor words.
Recognition of emotional words. | 24 hours after ketamine infusion
  Reaction time to categorise positive and negative descriptor words.
Recall of emotional words. | 24 hours after ketamine infusion
  Number of words correctly (hits) and incorrectly (false alarms) recalled.

CONTACTS AND LOCATIONS:
Overall Officials: Catherine Harmer, PhD, Principal Investigator — University of Oxford
Locations (1):
- University of Oxford, Oxford, United Kingdom

IPD SHARING:
Plan to Share IPD: Undecided